CLINICAL TRIAL: NCT03851029
Title: Comparison of Aerobic & Tai Chi Exercise on Cardiopulmonary Endurance Levels Among the Smoker University Students
Brief Title: Aerobic and Tai Chi Exercise Among the Smoker University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RiphahIU Ibraheem Zafar
Record Dates: First submitted 2019-02-08; First posted 2019-02-22 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Smoking, Cigarette
Keywords: Aerobic Exercise; Smoking; Tai Chi Exercise; University Student
MeSH Terms: conditions — Cigarette Smoking; Smoking | interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai chi (Experimental): (Yang 24 postures) Moderate intensity HRR (40%-60%)
  Interventions: Other: Tai chi
- Aerobic Training (Active Comparator): Elliptical Moderate intensity HRR (40%-60%)
  Interventions: Other: Aerobic Training

INTERVENTIONS:
Other: Tai chi — Session:
  • 3 times a week for 30-45 min.
  Duration:
  • For 6 weeks
  Warm-up:
  • 10-15 mints
  Cool-down:
  • 10-15 mints or stretching's
  Exercises time:
  • 20-30 mints
  Arms: Tai chi
Other: Aerobic Training — Session:
  • 3 times a week for 30-45 min.
  Duration:
  • For 6 weeks
  Warm-up:
  • 10-15 mints
  Cool-down:
  • 10-15 mints or stretching's
  Exercises time:
  • 20-30 mints
  Arms: Aerobic Training

SUMMARY:
It has also been observed that exercise reduces weight gain up to two years after quitting. Weight gain is often mentioned as a reason not to quit smoking, or as a reason to start smoking again. In addition, exercise has many other general benefits for smokers who have quit. However, the focus of the current research is the evaluate the effect of Aerobic& Tai Chi exercise on cardiopulmonary endurance levels among the smoker students within the University of Lahore. On the basis of comparison between two techniques, the study further concludes the findings by highlighting the strength of each technique.

DETAILED DESCRIPTION:
Currently, in Latin America and in the world, there is a strong focus on treatment and prevention in the population of all ages, with an emphasis on identifying and reducing modifiable risk factors that increases the possibility of chronic disease development among smokers.

Due to limited knowledge, people have develop the conception that Tai-Chi is not effective as much as high intensity exercises such as hiking, jumping ropes, biking and other aerobic exercises. Since last three decades the controversy related to effectiveness of Tai-chi exercises was persistent and to avoid the confusion a research was conducted on 25 Tai-chi students age range between 20-60years. The students were enrolled in the course of 7 years and was learning Yang style of Tai chi. The researchers have selected blood pressure, pulse and heart rate to assess the effectiveness of Tai-chi techniques and the data was recorded before and after the training of Tai-chi techniques. Through the findings of the study, they have observed that with light or easy frequency, the heart rate out of the maximum heart rate, the cardiovascular stimulus reached between 60 to 80% of the criteria introduced by the American Heart Association (AHA).

Accordingly, if these exercises performed at high performance, there was a minimum stimulation of the heart and observed at less than 60% of the maximum heart rate. Therefore, people who suffer from high blood pressure, or those who recovered from heart attacks or heart surgeries, high performance is a better option. According to specialists, a person can easily reach the standards set by the AHA by practicing Tai Chi three times a day.

When Tai Chi movements are performed quickly, they have the same beneficial effect on the cardiovascular system as aerobic exercise without creating the tension or stress. The physical stimulation can the be achieved by practicing the slow movements while using weights on the ankles, arms or body. Tai Chi is a very safe way of doing exercises and offers the same benefits as aerobic exercises, with no subsequent consequences.

Researchers state that high intensity exercise cannot be considered a complete physical activity. Although their influence on cardiovascular and muscular disorders is very high, but they do not necessary benefit other part of the body. On the other hand, Tai Chi has a significant impact on the overall body system and has the ability to rehabilitate any kind of body functioning disorder as compared to aerobic exercises. Along with that, age limitation, muscle strength and other environmental factors are the major concerns that influence the ability of performing Aerobic exercises with the full capacity. However, this is not the case with Tai-Chi exercises, in fact clinicians advise older people to perform the Tai chi technique to reduce the effect of cardiac disorders and improve body immune system.

On the other hand, traditional and advanced medical treatment, physical activity and exercise in the form of aerobic exercises are well-organized therapies for Heart failure risks. Although, researchers have presented controversial arguments related to the effectiveness of aerobic exercises with respect to rehabilitation, and continuous practice of such technique has shown quite positive and admirable effects to improve cardiac function, and reduced symptoms related to HF. In people with normal cardiac function, the practice of aerobic exercise results in a better cardiovascular function and better oxygen consumption as well as a lower heart rate at rest and a greater double product. The improvement in oxygen consumption is the result of an increase in cardiac performance and a greater extraction of oxygen in the muscles that are working. The best cardiac performance results from an increase in ventricular filling and beat volume.

Most importantly, Taichi not only supposes a multitude of advantages in the systems and parts of the body that habitually can improve with other exercises, but also it affects the circulation of the blood and the arterial tension because it activates intestinal functioning of the nervous system. Each of the movements of Tai Chi seeks to channel and release all energy to achieve a state of maximum peace of mind. In order to achieve the desired effects, concentration is extensively important along with breathing and movements.

ELIGIBILITY:
Inclusion Criteria:

* University students of smokers (Mild to moderate) (nicotine level)

Exclusion Criteria:

* Person with psychiatric disorders, neurological disorders, malignancies.
* Diagnosed Cardiac disease.
* Age less than 18 years and more than 27 years.
* Musculoskeletal disease that he was unable to perform aerobic exercises,
* Neuromuscular diseases that he was unable to maintain balance,
* Pulmonary issues like asthmatic students will be excluded

Ages: 18 Years to 27 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — smoking in our society female do not disclose or unwilling to participate in research even with consent
Enrollment: 87 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Shuttle run test (VO2 max) | 6 weeks
  Changes from the Baseline. This test is used to measure cardiopulmonary and cardiovascular fitness and maximum oxygen uptake VO2 max. VO2 max= 3.46*(L+SN/ (L*0.4325+7.0048)) + 12.2) Rating from Excellent to Poor cardiopulmonary endurance.

SECONDARY OUTCOMES:
Nicotine (cotinine drug test kit) urine strip tests: | 6 weeks
  Changes from the Baseline. The actual level of impregnation can be found more accurately by assessing the concentration of cotinine in the urine according to 3 detection levels (low / medium / high). Low concentration 1-3 cigarettes per day, Medium 3 to 10 cigarettes per day and High concentration 10 cigarettes per day
Digital Spirometer peak expiratory flow PEF, FEV1 - Forced Expiratory Volume and Forced vital Capacity FVC | 6 weeks
  Changes from the Baseline. The digital spirometer is used in clinical setting to analyze peak expiratory flow PEF in Liter/second. FEV1 - Forced Expiratory Volume in One Second in liter and Forced vital Capacity in Liter
Glover Nilsson Smoking Behavioral Questionnaire (GN-SBQ) | 6 weeks
  Changes from the baseline The Glover-Nilsson Smoking Behavior Questionnaire (GN-SBQ) is a self-report measure of behavioral dependence based on behaviors that may surround smoking or thoughts about smoking. Scores fall within a range of 0-33, with scores of 0 indicating mild behavioral dependence, and scores of 33 indicating very strong behavioral dependence

CONTACTS AND LOCATIONS:
Overall Officials: Sumaiyah Obaid Baig, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pleis JR, Ward BW, Lucas JW. Summary health statistics for U.S. adults: National Health Interview Survey, 2009. Vital Health Stat 10. 2010 Dec;(249):1-207. PMID 21905346
- [Background] Nelson ME, Rejeski WJ, Blair SN, Duncan PW, Judge JO, King AC, Macera CA, Castaneda-Sceppa C; American College of Sports Medicine; American Heart Association. Physical activity and public health in older adults: recommendation from the American College of Sports Medicine and the American Heart Association. Circulation. 2007 Aug 28;116(9):1094-105. doi: 10.1161/CIRCULATIONAHA.107.185650. Epub 2007 Aug 1. PMID 17671236
- [Background] D'Agostino RB Sr, Vasan RS, Pencina MJ, Wolf PA, Cobain M, Massaro JM, Kannel WB. General cardiovascular risk profile for use in primary care: the Framingham Heart Study. Circulation. 2008 Feb 12;117(6):743-53. doi: 10.1161/CIRCULATIONAHA.107.699579. Epub 2008 Jan 22. PMID 18212285
- [Background] Kuramoto AM. Therapeutic benefits of Tai Chi exercise: research review. WMJ. 2006 Oct;105(7):42-6. PMID 17163086
- [Background] Nedeljkovic M, Ausfeld-Hafter B, Streitberger K, Seiler R, Wirtz PH. Taiji practice attenuates psychobiological stress reactivity--a randomized controlled trial in healthy subjects. Psychoneuroendocrinology. 2012 Aug;37(8):1171-80. doi: 10.1016/j.psyneuen.2011.12.007. Epub 2012 Jan 4. PMID 22222120
- [Background] Yeh GY, Wang C, Wayne PM, Phillips RS. The effect of tai chi exercise on blood pressure: a systematic review. Prev Cardiol. 2008 Spring;11(2):82-9. doi: 10.1111/j.1751-7141.2008.07565.x. PMID 18401235
- [Background] Taylor-Piliae RE, Silva E, Sheremeta SP. Tai Chi as an adjunct physical activity for adults aged 45 years and older enrolled in phase III cardiac rehabilitation. Eur J Cardiovasc Nurs. 2012 Mar;11(1):34-43. doi: 10.1016/j.ejcnurse.2010.11.001. PMID 21095159
- [Background] Barrow DE, Bedford A, Ives G, O'Toole L, Channer KS. An evaluation of the effects of Tai Chi Chuan and Chi Kung training in patients with symptomatic heart failure: a randomised controlled pilot study. Postgrad Med J. 2007 Nov;83(985):717-21. doi: 10.1136/pgmj.2007.061267. PMID 17989272
- [Background] Redwine LS, Tsuang M, Rusiewicz A, Pandzic I, Cammarata S, Rutledge T, Hong S, Linke S, Mills PJ. A pilot study exploring the effects of a 12-week t'ai chi intervention on somatic symptoms of depression in patients with heart failure. J Altern Complement Med. 2012 Aug;18(8):744-8. doi: 10.1089/acm.2011.0314. Epub 2012 Jul 30. PMID 22845485
- [Background] Taylor-Piliae RE, Froelicher ES. Effectiveness of Tai Chi exercise in improving aerobic capacity: a meta-analysis. J Cardiovasc Nurs. 2004 Jan-Feb;19(1):48-57. doi: 10.1097/00005082-200401000-00009. PMID 14994782
- [Background] Jones LW, Eves ND, Peterson BL, Garst J, Crawford J, West MJ, Mabe S, Harpole D, Kraus WE, Douglas PS. Safety and feasibility of aerobic training on cardiopulmonary function and quality of life in postsurgical nonsmall cell lung cancer patients: a pilot study. Cancer. 2008 Dec 15;113(12):3430-9. doi: 10.1002/cncr.23967. PMID 18988290
- [Background] Downing J, Balady GJ. The role of exercise training in heart failure. J Am Coll Cardiol. 2011 Aug 2;58(6):561-9. doi: 10.1016/j.jacc.2011.04.020. PMID 21798416
- [Background] Moholdt TT, Amundsen BH, Rustad LA, Wahba A, Lovo KT, Gullikstad LR, Bye A, Skogvoll E, Wisloff U, Slordahl SA. Aerobic interval training versus continuous moderate exercise after coronary artery bypass surgery: a randomized study of cardiovascular effects and quality of life. Am Heart J. 2009 Dec;158(6):1031-7. doi: 10.1016/j.ahj.2009.10.003. PMID 19958872